CLINICAL TRIAL: NCT01103908
Title: Ultrasound Dilution Cardiac Output at the Conclusion of Cardiopulmonary Bypass in Pediatric Patients
Brief Title: Cardiac Output Measurement at the Conclusion of Cardiopulmonary Bypass
Status: Terminated | Type: Observational
Why Stopped: Site PI left position and lack of a suitable replacement PI.
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-G-HCE101-5A-H; 2R44HL082022-02 (NIH)
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Cardiac Output
Keywords: cardiac output; cardiopulmonary bypass; ultrasound dilution

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric cardiac output (CO) after CPB: Cardiac output measurements made in pediatric patients after cardiopulmonary bypass.
  Interventions: Device: HCE101 Cardiopulmonary Support Monitor

INTERVENTIONS:
Device: HCE101 Cardiopulmonary Support Monitor — Measurement of cardiac output using ultrasound dilution technology. The ultrasound dilution technology is in the HCE101 Cardiopulmonary Support Monitor.

SUMMARY:
Cardiac output, the amount of blood pumped by the heart in one minute, will be measured in pediatric patients undergoing surgery involving cardiopulmonary bypass (CPB). Cardiac output will be measured after cardiopulmonary bypass using a device that employs ultrasound dilution technology. At times, cardiac output will be measured during a procedure called modified ultrafiltration (MUF). The ultrasound dilution cardiac output measurements will be validated or compared with cardiac output measurements made using other FDA approved techniques and devices.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (age < 21 years)
* Pediatric patients undergoing surgery involving cardiopulmonary bypass

Exclusion Criteria:

* Patients aged > 21 years
* Patients undergoing surgery "off pump" (not involving cardiopulmonary bypass)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cardiac output measurements made in pediatric patients after cardiopulmonary bypass.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Cardiac output after cardiopulmonary bypass | Less than 10 minutes
  Cardiac output will be measured in pediatric patients after undergoing surgery involving cardiopulmonary bypass

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai Krivitski, PhD, DSc, Principal Investigator — Transonic Systems Inc.; Alistair Phillips, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No